CLINICAL TRIAL: NCT01223625
Title: Effect of Intensive Lipid Lowering Treatment Compared to Moderate Lipid Lowering Treatment on Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Rasmus Egede, Department of Cardiology, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF-200600
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2007-07

CONDITIONS: Endothelial Dysfunction; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin 5mg/day (Active Comparator): Rosuvastatin 5mg/day
  Interventions: Drug: Rosuvastatin 5mg/day
- Rosuvastatin 40mg/day (Active Comparator): Rosuvastatin 40mg/day
  Interventions: Drug: Rosuvastatin 40mg/day

INTERVENTIONS:
Drug: Rosuvastatin 5mg/day — Rosuvastatin 5mg/day
  Other Names: Crestor
  Arms: Rosuvastatin 5mg/day
Drug: Rosuvastatin 40mg/day — Rosuvastatin 40mg/day
  Other Names: Crestor
  Arms: Rosuvastatin 40mg/day

SUMMARY:
The aim of this study was to measure the effect of moderate and intensive lipid-lowering treatment with rosuvastatin on the endothelial function.

ELIGIBILITY:
Inclusion Criteria:

1. STEMI
2. no prior treatment with statins

Exclusion Criteria:

1. age below 18 or above 81 years
2. unconscious patients
3. serum creatinine > 176μmol/L
4. total-cholesterol > 7.0 mmol/l
5. hypothyreoidism ((TSH > 1.5 x ULN (upper limit of normal))
6. current liver disease (ALAT > 2 x ULN)
7. unexplained creatine kinase > 3 x ULN
8. alcohol or drug abuse within the last five years
9. prior myopathy or serious hypersensitivity reaction caused by statins
10. women with childbearing potential who were not using chemical or mechanical contraception
11. pregnant or breastfeeding women
12. history of malignancy unless a disease-free period of more than five years was present
13. patients with abnormal lung function test (LFT)
14. participation in another investigational drug study less than four weeks before enrolment in the present study
15. treatment with cyclosporine or fibrates.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The change from baseline in endothelium-dependent flow mediated vasodilatation of the brachial artery. | One year

SECONDARY OUTCOMES:
The change from baseline in endothelium independent flow mediated vasodilatation of the brachial artery | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Egede, MD, Principal Investigator — Department of Cardiology, Odense University Hospital, Odense, Denmark.
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Fuenen, Denmark

REFERENCES:
- [Derived] Egede R, Jensen LO, Hansen HS, Antonsen L, Hansen KN, Junker A, Thayssen P. Effect of intensive lipid-lowering treatment compared to moderate lipid-lowering treatment with rosuvastatin on endothelial function in high risk patients. Int J Cardiol. 2012 Jul 26;158(3):376-9. doi: 10.1016/j.ijcard.2011.01.071. Epub 2011 Feb 23. PMID 21349594